CLINICAL TRIAL: NCT00994591
Title: Cotinine Metabolism in Infants and Children
Acronym: 1058
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-03693
Record Dates: First submitted 2009-10-06; First posted 2009-10-14 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Secondhand Smoke Exposure
Keywords: Nicotine; Cotinine; CYP2A6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacokinetic dosing (Experimental)
  Interventions: Drug: Pharmacokinetic dosing

INTERVENTIONS:
Drug: Pharmacokinetic dosing — Pharmacokinetic testing involves dosing with deuterated cotinine which has an associated IND#61329.

SUMMARY:
Levels of cotinine, a biomarker for nicotine, have been found to be higher in infants and small children than adults. This pharmacokinetic study is designed to determine whether children metabolize cotinine differently than adults.

Seventy-two healthy children between the ages of 2 months and 6 years will come with their mothers to SFGH GCRC for one approximately 9 hour visit. After being examined by a pediatrician, the child will be administered one dose of cotinine at .05 mg/kg.

Saliva and urine samples will be collected prior to dosing and throughout the day to characterize the metabolism and excretion of cotinine. The investigators have previously shown that a ratio of 3'-hydroxycotinine/cotinine (3HC/Cot) in saliva correlates closely to nicotine metabolism.

Following these one day hospital visits, a research assistant will visit the participants in their homes to collect urine and saliva samples at 1,2,3,7, and 10 days after the initial dose.

DETAILED DESCRIPTION:
The long-term goal is to characterize developmental changes in CYP2A6 activity and nicotine and cotinine metabolism in infants and children. Our hypotheses are:

* The rate of nicotine and cotinine metabolism and the level of CYP2A6 activity will increase with age throughout infancy and childhood.
* The rate of cotinine glucuronidation (reflecting UGT 1A4 and 1A9 activity) will increase with age.
* Cotinine clearance will be lower and cotinine half-life longer in African-Americans compared to Caucasians.
* The excretion of cotinine glucuronide will be less among African-Americans compared to Caucasians.
* Developmental increases in CYP2A6 will be greatest in children with wild type CYP2A6 genes, and will be lower in children who have CYP2A6 gene variants associated with reduced activity.

This present study is the first step in the investigation of the above hypotheses. The primary goal of this study is to determine if there are age-related changes in cotinine clearance and validate the 3HC/COT ratio as a biomarker of cotinine clearance and half-life. This biomarker can then be used in larger studies to explore the hypotheses described above. The biomarker could also be used in epidemiologic studies of the health effects of SHS in infants and children.

Primary Specific Aims:

1. Determine the following in infants and children between 2 and 84 months of age dosed with deuterium-labeled cotinine:

   * The clearance of cotinine
   * The half-life of cotinine
   * The volume of distribution of cotinine
2. Validate the 3HC/Cot ratio in saliva and in urine as a marker of cotinine clearance and half-life.

   Secondary Specific Aims:
3. Determine the effects of age on the cotinine metabolite profile in the 8-hour urine sample.
4. Determine if sulfation is a conjugation pathway for cotinine in infants and young children.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 12 months, 13-24 months, and 25-83 months
* Caucasian (including Hispanic) and African American only
* Some exposure to secondhand smoke

Exclusion Criteria:

* Any medical problems
* Taking prescription medication (there are exceptions)

Ages: 2 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Cotinine clearance | 8 hours

SECONDARY OUTCOMES:
Half-life of cotinine | 8 hour

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, SFGH, CTSI,CRC, San Francisco, California, United States